CLINICAL TRIAL: NCT05095935
Title: Medtronic Signia Small Diameter Reload Product Surveillance Registry
Brief Title: Medtronic Signia SDR Product Surveillance Registry
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Surgical PSR
Record Dates: First submitted 2021-08-24; First posted 2021-10-27 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2024-10

CONDITIONS: Minimally Invasive Surgical Procedures; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Thoracic Adult: Use of Signia SDR for the transection of pulmonary arteries and veins in adult patients.
  Interventions: Other: N/A observational registry
- Abdominal Adult: Use of Signia SDR for the transection of renal arteries and veins in adult patients.
  Interventions: Other: N/A observational registry
- Abdominal Pediatric: Use of Signia SDR for the transection of the appendiceal stump and mesoappendix (simple acute appendicitis) in pediatric patients.
  Interventions: Other: N/A observational registry

INTERVENTIONS:
Other: N/A observational registry — N/A observational registry

SUMMARY:
The purpose of the registry is to confirm the safety and performance of the Signia™ Small Diameter Reload (SDR) when used in surgical procedures in a real-world setting in patients receiving surgery for indicated thoracic, abdominal, and pediatric applications, intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements
* Patient has, or is intended to receive or be treated with, an eligible Medtronic product
* Patient is consented within the enrollment window of the therapy received, as applicable

Exclusion Criteria:

* Patient who is, or is expected to be, inaccessible for follow-up
* Patient is excluded by local law
* Patient is currently enrolled in, or plans to enroll in, any concurrent drug/device study that may confound the PSR results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgical procedures during which the Signia Small Diameter Reload is being used for transection of the arteries and veins meeting the cohort criteria.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Children's Hospital Colorado, Denver, Colorado
  - The George Washington University Hospital, Washington D.C., District of Columbia
  - Rush, Chicago, Illinois
  - Cooper Health System, Camden, New Jersey
  - NYU Langone Medical Center, New York, New York
  - New York Presbyterian Hospital - Colombia University Medical Center, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health Systems, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Falk Clinic, Pittsburgh, Pennsylvania
  - University of Texas - San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Mary Washington Hopital, Fredericksburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing surgical procedures during which the Signia Small Diameter Reload is being used for the transection of vasculature or thin tissue meeting the cohort criteria were considered for this study.
Pre-assignment Details: This study was conducted in accordance with each site's standard of care. Assignment to one of the three study groups was dependent on the anatomical location where Signia SDR was used and was not randomly assigned.
Period: Overall Study
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Started | 123 | 163 | 95
Completed | 123 | 163 | 95
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 430 subjects were enrolled in the study, however, 49 subjects ultimately were not treated with Signia SDR and as such they were considered screen failures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric | Total
Number analyzed (Participants) | 123 | 163 | 95 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (12.1) | 48.4 (13.5) | 11.3 (3.8) | 44.9 (23.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 95 | 31 | 192
  Male | 57 | 68 | 64 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 20 | 42 | 67
  Not Hispanic or Latino | 109 | 130 | 53 | 292
  Unknown or Not Reported | 9 | 13 | 0 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 3 | 5 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 28 | 10 | 44
  White | 107 | 100 | 49 | 256
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 6 | 27 | 33 | 66
Region of Enrollment [Number; unit: Participants]
  United States | 123 | 163 | 95 | 381

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Intraoperative Hemostatic Intervention
Description: * Adult Thoracic: incidence of intraoperative hemostatic intervention related to the transection of pulmonary arteries and veins.
  * Adult Abdominal: incidence of intraoperative hemostatic intervention related to the transection of renal arteries and veins.
  * Pediatric Abdominal: incidence of intraoperative hemostatic and leak intervention related to the transection of the appendiceal stump and mesoappendix (simple acute appendicitis).
Time Frame: During Procedure
Population: Analysis was conducted on the number of firings of the Signia SDR device. Study participants could have 1 or more firings.
Measure: Count of Units; unit: Firings
Units Other Than Participants: Firings
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 123 | 163 | 95
Number analyzed (Firings) | 302 | 327 | 100
Firings | 3 | 2 | 0

2. Secondary Outcome: Incidence of Repeat Hospital Admission for Primary Procedure-related Complications
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 120 | 157 | 95
Participants | 1 | 1 | 0

3. Secondary Outcome: Intraoperative Assessments: Assessment of Staple Line Integrity Using a Five-point Likert Scale
Description: The Likert Scale assessment is a bleeding assessment that was conducted during the procedure, ranging from 1 (no bleeding) to 5 (significant bleeding requiring intervention). Staple line integrity was considered achieved for firings with a Likert Scale Score of 1, 2, 3 and 777 (not recorded at time of procedure, but deemed acceptable by the procedure surgeon).
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 120 | 157 | 95
Participants | 117 | 156 | 95

4. Secondary Outcome: Intraoperative Assessments: Incidence of Staple Line Bleeding
Description: Number of firings that had an incidence of staple line bleeding of >50cc
Time Frame: During Procedure
Measure: Count of Units; unit: Firings
Units Other Than Participants: Firings
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 120 | 157 | 95
Number analyzed (Firings) | 302 | 327 | 100
Firings | 0 | 0 | 0

5. Secondary Outcome: Intraoperative Assessments: Additional Intervention(s) to Treat Staple Line Failure
Description: Additional interoperative interventions to treat staple line failure (applying additional stapler reloads, applying compression greater than what is considered typical, over-sewing with suture, placing clips, use of energy, use of seatbelt, other)
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 120 | 157 | 95
Participants | 3 | 1 | 0

6. Secondary Outcome: Post-operative Assessments: Additional Intervention(s) to Treat Staple-line Failure
Description: Additional postoperative interventions to treat staple line failure (Applying additional stapler reloads, Applying compression greater than what is considered typical, Over-sewing with suture, Placing clips, Use of energy, Use of seatbelt, Other)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 120 | 157 | 95
Participants | 0 | 0 | 0

7. Secondary Outcome: Device Deficiencies
Description: incidence of subjects reporting device deficiencies affecting the intended performance of the device up to and including 30 days following the use of device (i.e. Signia™ Small Diameter Reloads) in surgery
Time Frame: 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
Number analyzed (Participants) | 123 | 163 | 95
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: from enrollment until end of 30 day follow-up
Description: Procedure and/or device related AEs were reportable in this study. Subject follow-up period was 30-days post procedure; no events were collected beyond 30-days post procedure.
Arm/Group | Thoracic Adult | Abdominal Adult | Abdominal Pediatric
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/163 | 0/95
Serious Adverse Events (participants affected / at risk) | 43/123 | 7/163 | 4/95
Other Adverse Events (participants affected / at risk) | 6/123 | 6/163 | 8/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic Adult (N=123) | Abdominal Adult (N=163) | Abdominal Pediatric (N=95)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 24 (24) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 10 (10) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drug Intolerance (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Burkholderia Cepacia Complex Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia Acinetobacter (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 10 (10) | 0 (0) | 0 (0)
Pneumonia Escherichia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Fungal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia Klebsiella (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia Pseudomonal (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 7 (8) | 0 (0) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Stenotrophomonas Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Streptococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Systemic Candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vasoplegia Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Device Leakage (Product issues) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic Adult (N=123) | Abdominal Adult (N=163) | Abdominal Pediatric (N=95)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Adverse Drug Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy To Surgical Sutures (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Incision Site Discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Constipation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Device Leakage (Product Issues) | 2 (2) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish as long as publications are provided to Medtronic for review at least 30 days prior to submission or presentation. Additionally, PIs will not independently publish, publicly disclose, present or discuss any Study results until a multi-center publication is released. If a multi-center publication is not released within one year after completion PIs will have the right to publish the results of and information pertaining to their activities on the Study.

DOCUMENTS (2):
  • Study Protocol (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT05095935/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT05095935/SAP_001.pdf